CLINICAL TRIAL: NCT02258100
Title: Retrospective Review of an Anesthesia Information System and Paper Anesthesia Records for Care Congruency in a Single Surgical Population.
Brief Title: Anesthesia Information System vs Paper Anesthesia Records for Care Congruency
Status: Completed | Type: Observational
Sponsor: Endeavor Health (Other)
Responsible Party: Sponsor
Other Study IDs: EH14-325
Record Dates: First submitted 2014-10-01; First posted 2014-10-07 (Estimated); Last update posted 2019-09-11 (Actual); Status verified 2019-09

CONDITIONS: Paper Versus EMR Generated Anesthesia Records
MeSH Terms: interventions — Electronic Health Records

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Paper: Patients receiving care documented via paper anesthesia record.
- AIMS: Patients receiving care documented via electronic anesthesia record.
  Interventions: Other: Electronic Medical Record

INTERVENTIONS:
Other: Electronic Medical Record — Advent of EMR use for documentation of anesthetic care
  Groups: AIMS

SUMMARY:
To date the effect of AIMS on medical interventions has not been studied. We seek to retrospectively evaluate paper and electronic anesthesia records among a single surgical population (esophageal surgery) to ascertain any differences that may exist between cohorts with regards to chart completion, anesthetic management and medical care.

DETAILED DESCRIPTION:
Anesthesia information systems (AIMS) are increasingly used to electronically capture physiologic and management data during anesthesia. Proponents tout an improved accuracy of data yet this has not been formally evaluated. Furthermore, whether AIMS is associated with changes in medical care is unknown. Studies with newer technologies have demonstrated increased medical interventions as a result of implementation. The pulmonary artery catheter was shown to increase medical interventions when used yet no improvement in outcomes are observed and some suggest a deleterious effect. 1 Several studies suggest improved patient care with electronic anesthesia records. 2,3 These all center around clinical decision support that reminds clinicians to give certain medications or ensure chart completion. Despite these advantages there are no studies evaluating the 'hawthorne effect' of AIMS. Physiologic data is now recorded at each data point using AIMS. This differs significantly from paper anesthesia records in which clinicians often chart physiologic trends choosing to omit spurious values. It is possible that a Hawthorne effect may occur in this scenario with increased data collection and an increased ability to scrutinize the medical record. Given the litigious nature of medical practice today, there is concern about the impact of AIMS on medicolegal liability. 4 Yet, to date the effect of AIMS on medical interventions has not been studied. We seek to retrospectively evaluate paper and electronic anesthesia records among a single surgical population (esophageal surgery) to ascertain any differences that may exist between cohorts with regards to chart completion, anesthetic management and medical care.

ELIGIBILITY:
Inclusion Criteria:

* Underwent esophageal surgery and had anesthetic documented in medical record

Exclusion Criteria:

* Cases less than one hour

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who underwent esophageal surgery with one surgeon from 2009-2014
Sampling Method: Non-Probability Sample
Enrollment: 189 (Actual)
Dates: Start 2014-09; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Anesthetic Care; Drugs delivered | Anesthesia start to Anesthesia Stop
  Intraoperative anesthetic medications; Total dose and number of interventions for all drugs; Fentanyl, ephedrine, phenylephrine, norepinephrine, labetalol, nicardidipine, esmolol, hydrazine
documented hypotension | Anesthesia start to Anesthesia End (Intraoperative)
  Intraoperative hypotension; Each occurrence less then 20% of patient's baseline, calculated from preoperative systolic BP; Duration of hypotension; associated medical treatment

CONTACTS AND LOCATIONS:
Overall Officials: Torin D Shear, MD, Principal Investigator — Endeavor Health
Locations (1):
- Evanston Hospital, Evanston, Illinois, United States